CLINICAL TRIAL: NCT02292108
Title: Study of the Influence of Erickson's Hypnosis and Self-hypnosis Practice on Food Impulsivity and Weight Loss in Obese Patients: a Pilot Project
Brief Title: Hypnosis, Self-hypnosis and Weight Loss in Obese Patients
Acronym: HYPNODIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P131202
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2017-01

CONDITIONS: Obesity
Keywords: Hypnosis; self-hypnosis; obesity; high food impulsiveness
MeSH Terms: conditions — Obesity | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis and dietetic counselling (Experimental): Patient will benefit of usual dietetic counselling and experimental hypnosis
  Interventions: Behavioral: dietetic counselling; Behavioral: Hypnosis and self-hypnosis
- dietetic counselling (Other): Patient will only benefit of usual dietetic counselling
  Interventions: Behavioral: dietetic counselling

INTERVENTIONS:
Behavioral: dietetic counselling
Behavioral: Hypnosis and self-hypnosis — Erickson's hypnosis and self-hypnosis
  Arms: Hypnosis and dietetic counselling

SUMMARY:
High food impulsiveness, impaired food reward and stress response are involved in the phenomena of weight gain and resistance at weight loss. Henceforth, hypnosis is a complementary medicine which is recognized as effective for defined indications. Complexity and diversity of methodological studies with hypnosis does not allow to conclude on its efficacy in treating this disease.

In obese subjects with high food impulsiveness, it is expected that Erickson's hypnosis and self-hypnosis practice would improve food disinhibition assessed by an adapted questionary (TFEQ 51).

DETAILED DESCRIPTION:
Obese failing patients are recruited in an university hospital. Half of the subjects will be randomised to practice hypnosis and will learn to practice self-hypnosis to reduce food impulsivity and specially disinhibition. In the same time, all the included patients will follow therapeutic workshops based on current recommendations of the High Health Authority of France (HAS) for physical activity and the dietetic.

In the hypnosis group, eight workshops are planned during six months. Furthermore, patients have to practice daily self-hypnosis. In the same time, all the patients included will participate in eight dietetic workshops.

It is expected an improvement in patient involvement in personalized care plan, that eating behavior is more suited and consequently a significant decrease in weight.

ELIGIBILITY:
Inclusion criteria :

* subjects adult volunteers under 70 years old
* high score of disinhibition (D> 8)
* obesity grade 1 and 2 (BMI between 30 and 40 kg m ²)
* no previous practice of hypnosis

Exclusion criteria :

* weight change of more than 3 kg peak to peak in the last 6 months
* psychiatric illness known
* craniopharyngioma
* treatment with a significant influence on the weight and / or eating behavior: steroids, hyperthyroidism, uncontrolled hypothyroidism,
* bariatric Surgery
* major TCA according to DSM IV
* sensory impairments (hearing, visual skills) and cognitive impairing its award of rating scales
* planned or ongoing pregnancy
* refusal of hypnosis.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Evolution of disinhibition score estimated by the TFEQ 51 at the beginning and at the end of the study | 8 months

SECONDARY OUTCOMES:
Evolution of cognitive restraint at the beginning and at the end of the study | 8 months
  Cognitive restraint estimated by the Three Factor Eating Questionnaire (TFEQ 51)
Evolution of flexible cognitive restraint at the beginning and at the end of the study | 8 months
  Flexible cognitive restraint estimated by the Three Factor Eating Questionnaire (TFEQ 51)
Evolution of rigid cognitive restraint at the beginning and at the end of the study | 8 months
  Rigid cognitive restraint estimated by the Three Factor Eating Questionnaire (TFEQ 51)
Evolution of weight at the beginning and at the end of study | 8 months
  Weight will be measured in Kg
Evolution of waist circumference at the beginning and at the end of study | 8 months
  Waist circumference will be measured in Cm
Evolution of body fat at the beginning and at the end of the study | 8 months
  Body fat will be measured in Kg using dual-energy X-ray absorptiometry (DXA)
Evolution of lean mass at the beginning and at the end of the study | 8 months
  Lean mass will be measured in Kg using dual-energy X-ray absorptiometry (DXA)
Evolution of water mass at the beginning and at the end of the study | 8 months
  Water mass will be measured in Kg using dual-energy X-ray absorptiometry (DXA)
Evolution of calories intakes. at the beginning and at the end of the study | 8 months
  calories will be measured in Kcal/day, assessed for 3 representative days (two weekdays and one weekend day) and collected using an interactive self-administered food journal from the internet enabled during the week prior to the inclusion visit and the final visit
Evolution of protein intakes.at the beginning and at the end of the study | 8 months
  Protein will be measured in g/day assessed for 3 representative days (two weekdays and one weekend day) and collected using an interactive self-administered food journal frome the internet enabled during the week prior to the inclusion visit and the final visit.
Evolution of carbohydrate intakes | 8 months
  carbohydrates be measured in g/day, assessed for 3 representative days (two weekdays and one weekend day) and collected using an interactive self-administered food journal from the internet enabled during the week prior to the inclusion visit and the final visit
Evolution of total fat intakes at the beginning and at the end of the study. | 8 months
  Total fat will be measured in g/day assessed for 3 representative days (two weekdays and one weekend day) and collected using an interactive self-administered food journal from the internet enabled during the week prior to the inclusion visit and the final visit
Evolution of saturated fatty acids intakes at the beginning and at the end of the study. | 8 months
  Saturated fatty acids will be measured in g/day assessed for 3 representative days (two weekdays and one weekend day) and collected using an interactive self-administered food journal from the internet enabled during the week prior to the inclusion visit and the final visit
Evolution of Total cholesterol at the beginning and the end of the study | 8 months
  Total cholesterol will be measured in g/L
Evolution of High-density lipoprotein-cholesterol (HDL-C) at the beginning and the end of the study | 8 months
  High-density lipoprotein-cholesterol (HDL-C) will be measured in g/L
Evolution of Low-density lipoprotein (LDL-C) at the beginning and the end of the study | 8 months
  Low-density lipoprotein (LDL-C) will be measured in g/L
Evolution of Triglyceride at the beginning and the end of the study | 8 months
  Triglyceride will be measured in g/L
Evolution of fasting glucose at the beginning and the end of the study | 8 months
  Fasting glucose will be measured in mmol/L
Evolution of HbA1c at the beginning and the end of the study | 8 months
  HbA1c will be measured in %
Evolution of quality of Live (QoL) estimated by The Short-Form Health Survey (SF-36) at beginning and the end of study at the beginning and the end of the study | 8 months
  Scores range from 0 to 100 with a higher score indicating a greater QoL.
Evolution of stress measured at beginning and the end of study. | 8 months
  stress will be measured by General Health Questionnaire (GHQ28)
Evolution of coping strategies measured by The Coping Inventory for Stressful Situations (CISS) at beginning and the end of study | 8 months
  In the Coping Inventory for Stressful Situations (CISS) items are scored on a 5-point Likert scale (from 1 not at all to 5 very much). Scores for all items per scale are summed to form scale scores; higher scores indicate a greater use of that coping strategy.
Evolution of the Self-esteem measured by The Self-esteem Inventory (SEI of Coopersmith) at beginning and the end of study | 8 months
  The Self-esteem Inventory (SEI of Coopersmith) consists of 58 items and 4 subscales: general, social, family and professional self-esteem. A lie score is also computed to capture social desirability in participants answers. Higher scores indicate a greater self-esteem..
: Evolution of the patient's involvement in the personalized care project evaluated by content analysis of a psychological interview at beginning and the end of study | 8 months
  Analysis of speech content using Sphinx software
: Evolution of the patient's emotional state evaluated by content analysis of a psychological interview at beginning and the end of study | 8 months
  Analysis of speech content using Sphinx software
Evolution of the food reward evaluated by content analysis of a psychological interview at beginning and the end of study | 8 months
  Analysis of speech content using Sphinx software
Evolution of the self-perception of self-care competence evaluated by content analysis of a psychological interview at beginning and the end of study | 8 months
  Analysis of speech content using Sphinx software
Evolution of the physical activity assessed with the abridged version of the International Physical Activity Questionnaire (IPAQ) completed online before the inclusion visit and before the final visit | 8 months
  In the abridged version of the International Physical Activity Questionnaire (IPAQ) walking, moderate Physical activity and vigorous Physical activity will be measure in min/week, the Sedentary will be measure in min/day
Evolution of the physical activity assessed with a pedometer for a week prior to the second and final visits. | 8 months
  Walking will be measure in number of steps/day

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Giral, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpetriere Hospital, Paris, France

REFERENCES:
- [Derived] Delestre F, Lehericey G, Estellat C, Diallo MH, Hansel B, Giral P. Hypnosis reduces food impulsivity in patients with obesity and high levels of disinhibition: HYPNODIET randomized controlled clinical trial. Am J Clin Nutr. 2022 Jun 7;115(6):1637-1645. doi: 10.1093/ajcn/nqac046. PMID 35170724